CLINICAL TRIAL: NCT05029713
Title: Sarcopenic Obesity and Associated Risk Factors in Patients Undergone Liver Transplant
Brief Title: Sarcopenic Obesity in Liver Transplanted Patients
Acronym: OSaLT
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Collaborators: Prof. Maria Grano (Unknown)
Responsible Party: Principal Investigator, Michele Barone, Associate Professor, University of Bari
Other Study IDs: Policlinico 8
Record Dates: First submitted 2021-07-17; First posted 2021-08-31 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Sarcopenic Obesity
Keywords: liver transplantation; obesity; sarcopenia; calcineurin inhibitors
MeSH Terms: conditions — Obesity; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- liver transplanted patients without sarcopenic obesity (controls): All liver transplanted patients followed as outpatients at out clinic, which lack at least one of the two conditions (muscle strenght and muscle mass) used to identify sarcopenic obesity.
  Interventions: Diagnostic Test: Evaluation of appendicular skeletal muscle mass (ASMM) by bioelectrical impedance analysis (BIA)
- liver transplanted patients with sarcopenic obesity (cases): All liver transplanted patients followed as outpatients at out clinic, with both muscle strenght and muscle mass.
  Interventions: Diagnostic Test: Evaluation of appendicular skeletal muscle mass (ASMM) by bioelectrical impedance analysis (BIA)

INTERVENTIONS:
Diagnostic Test: Evaluation of appendicular skeletal muscle mass (ASMM) by bioelectrical impedance analysis (BIA) — The use of handgrip dynamometer and BIA will be used to screen all liver transplanted patients for sarcopenic obesity, using a muscle strength cut-off <27 Kg in men and <16 Kg in women and a standardized muscle mass cut-off <0.789 ASMM/BMI for men and 0.512 ASMM/BMI for women.
  Other Names: Evaluation of muscle strenght by an handgrip dynamometer; Evaluation of physical activity by the International Physical Activity Questionnaire (IPAQ); The Yale Food Addiction Scale will be used to exclude risk of patients to binge

SUMMARY:
The prevalence of obesity in cirrhotic patients who are candidates for liver transplantation (LT) is increasing, a phenomenon consistent with the increased prevalence of obesity in the general population. On the other hand, in liver patients on the waiting list for transplantation it is often observed sarcopenia. The combination of the two condition is defined sarcopenic obesity, which combines the negative synergy deriving from the two conditions. In this study the investigators will evaluate, for the first time, the prevalence of sarcopenic obesity in subjects undergone LT and determine the possible associated risk factors, particularly the role of immunosuppressive treatment with calcineurin inhibitors in addition to dietary habits and physical activity.

DETAILED DESCRIPTION:
Obesity is a clinical condition characterized by excessive body weight due to the accumulation of adipose tissue, which represents a risk to health. In particular, obesity represents a risk factor for cardiovascular diseases, metabolic syndrome, NAFLD, and significantly increases the risk of mortality compared to normal weight subjects. It has been reported that the presence of obesity represents a risk factor for post-operative complications in patients undergone LT, increasing the mortality risk in those with the highest degree of obesity. At the same time, an evaluation obesity on the basis of body mass index (BMI) does not take in account the real body composition in terms of fat mass and muscle mass, which are more effective prognostic factors. Data of the literature report that patients undergoing liver transplantation (LT) have an average weight gain of 9 kg during the first year following the transplant, whereas in the second year, it would be observed about 24% incidence of obesity that would reach 30-38% in the third year. However, in all these studies the evaluation of de novo obesity is biased by the lack of data on the body weight of the patients prior their inclusion in the waiting list or to the use of dry body weight in patients mostly decompensated, or the loss of patients at the follow up. On the other hand, in liver patients on the waiting list for transplantation it is often observed sarcopenia, a syndrome characterized by progressive and generalized loss of skeletal muscle mass and strength associated with an increased risk of adverse events such as disability, poor quality of life and death. In this clinical setting, it has been reported in a percentage ranging from 41% to 68 %.

The combination of the two condition defined sarcopenic obesity, which combines the negative synergy deriving from the two conditions, has been reported to be 20-40% in patients on the waiting list for liver transplantation. In addition, calcineurin inhibitors, which represent the backbone of anti-rejection therapy, have been investigated for their negative effect on muscle mass.

In this study the investigators will evaluate, for the first time, the prevalence of sarcopenic obesity in subjects undergone LT and assess the possible associated risk factors, particularly the role of immunosuppressive treatment with calcineurin inhibitors (Ciclosporin and Tacrolimus), iin addition to dietary habits and physical activity. To achieve this goal the investigators will first screen all liver transplanted patients for muscle strenght and then all subjects with reduced muscle strenght will undergo bioelectrical impedance analysis (BIA). The presence of both conditions will allow us to identify subjects with sarcopenic obesity.

Finally, the immunosuppressive therapy will be compared in liver transplanted patients with and without sarcopenic obesity. The evaluation of risk factors for obesity will be completing by the assessment of dietary habits and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had a liver transplant for more than one year

Exclusion Criteria:

* patients who have had a liver transplant for less than one year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All liver transplanted patients who have had a liver transplant for more than one year
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Sarcopenic obesity prevalence in liver transplanted patients | At enrollment
  In all obese patients identified by a body mass index (BMI) ≥ 30 the investigators will first evaluate muscle strenght and those subjects with a reduction of muscle strenght (muscle strength <27 Kg in men and <16 Kg in women) will undergo the evaluation of muscle mass by bioelectrical impedance analysis; in the latter case the appendicular skeletal muscle mass (ASM) will be standardized for BMI (ASM/BMI), and the cut-offs considered will be <0.789 for men and <0.512 for women.

SECONDARY OUTCOMES:
The possible involvement of calcineurine inhibitors in patients with sarcopenic obesity | At enrollment
  The investigators will compare the prevalence of sarcopenic obesity in subjects receiving calcineurin with that observed in subjects receiving other therapies by the Chi squared or Fisher test. In case of a significantly different prevalence between the two groups, a multivariate analysis will be performed to confirm if calcineurin inhibitor therapy is an indipendent risk factor for sarcopenic obesity.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Policlinic Hospital, Bari, BA
  - Policlinic Hospital, Bari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barone M, Viggiani MT, Losurdo G, Principi M, Leandro G, Di Leo A. Systematic review with meta-analysis: post-operative complications and mortality risk in liver transplant candidates with obesity. Aliment Pharmacol Ther. 2017 Aug;46(3):236-245. doi: 10.1111/apt.14139. Epub 2017 May 10. PMID 28488418
- [Background] Barone M, Viggiani MT, Avolio AW, Iannone A, Rendina M, Di Leo A. Obesity as predictor of postoperative outcomes in liver transplant candidates: Review of the literature and future perspectives. Dig Liver Dis. 2017 Sep;49(9):957-966. doi: 10.1016/j.dld.2017.07.004. Epub 2017 Jul 22. PMID 28801180
- [Background] Rezende Anastacio L, Garcia Ferreira L, Costa Liboredo J, de Sena Ribeiro H, Soares Lima A, Garcia Vilela E, Correia MI. Overweight, obesity and weight gain up to three years after liver transplantation. Nutr Hosp. 2012 Jul-Aug;27(4):1351-6. doi: 10.3305/nh.2012.27.4.5768. PMID 23165585
- [Background] Everhart JE, Lombardero M, Lake JR, Wiesner RH, Zetterman RK, Hoofnagle JH. Weight change and obesity after liver transplantation: incidence and risk factors. Liver Transpl Surg. 1998 Jul;4(4):285-96. doi: 10.1002/lt.500040402. PMID 9649642
- [Background] Richards J, Gunson B, Johnson J, Neuberger J. Weight gain and obesity after liver transplantation. Transpl Int. 2005 Apr;18(4):461-6. doi: 10.1111/j.1432-2277.2004.00067.x. PMID 15773968
- [Background] Beckmann S, Nikolic N, Denhaerynck K, Binet I, Koller M, Boely E, De Geest S; Psychosocial Interest Group, Swiss Transplant Cohort Study. Evolution of body weight parameters up to 3 years after solid organ transplantation: The prospective Swiss Transplant Cohort Study. Clin Transplant. 2017 Mar;31(3). doi: 10.1111/ctr.12896. Epub 2017 Jan 24. PMID 28008650
- [Background] Hanai T, Shiraki M, Nishimura K, Ohnishi S, Imai K, Suetsugu A, Takai K, Shimizu M, Moriwaki H. Sarcopenia impairs prognosis of patients with liver cirrhosis. Nutrition. 2015 Jan;31(1):193-9. doi: 10.1016/j.nut.2014.07.005. Epub 2014 Jul 30. PMID 25441595
- [Background] Masuda T, Shirabe K, Ikegami T, Harimoto N, Yoshizumi T, Soejima Y, Uchiyama H, Ikeda T, Baba H, Maehara Y. Sarcopenia is a prognostic factor in living donor liver transplantation. Liver Transpl. 2014 Apr;20(4):401-7. doi: 10.1002/lt.23811. Epub 2014 Jan 27. PMID 24357065
- [Background] Schiavo L, Busetto L, Cesaretti M, Zelber-Sagi S, Deutsch L, Iannelli A. Nutritional issues in patients with obesity and cirrhosis. World J Gastroenterol. 2018 Aug 14;24(30):3330-3346. doi: 10.3748/wjg.v24.i30.3330. PMID 30122874
- [Background] Hudson MB, Price SR. Calcineurin: a poorly understood regulator of muscle mass. Int J Biochem Cell Biol. 2013 Oct;45(10):2173-8. doi: 10.1016/j.biocel.2013.06.029. Epub 2013 Jul 6. PMID 23838168